CLINICAL TRIAL: NCT02595346
Title: Efficiency of Hydroxychloroquine on the Endothelial Dysfunction in Antiphospholipid Syndrome (APLAQUINE)
Brief Title: Study of the Efficiency of Hydroxychloroquine on the Endothelial Dysfunction and Its Vascular Consequences During the Antiphospholipid Syndrome
Acronym: APLAQUINE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/074/HP
Record Dates: First submitted 2015-11-02; First posted 2015-11-03 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Antiphospholipid Syndrome (APS)
MeSH Terms: conditions — Antiphospholipid Syndrome | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- hydroxychlorquine (Experimental): hydroxychloroquine 200 mg twice a day for 6 months
  Interventions: Drug: Hydroxychloroquine
- control (Placebo Comparator): placebo 2 pills a day for 6 months
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — endothelial function is assessed by measuring the flow mediated dilatation of humeral artery in response to ischemia. the dilatation is evaluated by echotracking.
  glycocalyx thickness is measured by the study of sublingual microcirculation with SDF imaging.
  oxydative, inflammatory and coagulation parameters is assessed on plasma samples.
  Other Names: plaquenil
  Arms: hydroxychlorquine
Drug: placebo — endothelial function is assessed by measuring the flow mediated dilatation of humeral artery in response to ischemia. the dilatation is evaluated by echotracking.
  glycocalyx thickness is measured by the study of sublingual microcirculation with SDF imaging.
  oxydative, inflammatory and coagulation parameters is assessed on plasma samples.
  Arms: control

SUMMARY:
This study evaluates the benefits of hydroxychloroquine on arterial function in antiphospholipid syndrome.

Briefly, the patients will be randomized in two groups, one will receive hydroxychloroquine and standard treatment, the other will receive placebo in addition of standard treatment.

DETAILED DESCRIPTION:
Antiphospholipid syndrome (APS) is an autoimmune disease characterized by recurrent thrombotic events and miscarriages, with persistently positive antiphospholipid antibodies (aPL). APS may be isolated (primary APS) or associated to a connective tissue disease, most often systemic lupus erythematous (SLE).

Pathogenic effects of aPL were first described by the demonstration that in vitro incubation of endothelial cells or monocytes with aPL induce an endothelial dysfunction characterized by pro-coagulant (overexpression of tissue factor and modulation of protein C and S), pro-inflammatory (increased level of IL-6(interleukin 6) , IL-1β and TNFα) and pro-adhesive (increased levels of ICAM-1(intercellular adhesion molecule ), VCAM-1 (vascular endothelial cell adhesion molecule) and E-selectin) phenotypes. In parallel the investigators and others reported that endothelial function, assessed by flow mediated dilatation, is altered in patients with primary and secondary forms of APS. Although a role for TLR (toll-like receptor )-mediated NFkB translocation has been advanced, the pathogenic mechanisms that lead to in vivo endothelial injury in APS are incompletely understood.

In an experimental model, the investigators demonstrated that passive transfer of human aPL to mice induced a marked endothelial dysfunction assessed ex vivo in small resistance arteries, and an increase in TNFα levels. Moreover, the investigators group have demonstrated that patients with primary arterial APS display endothelial dysfunction and structural arterial changes, associated with a pro-oxidative and pro-coagulant state and with activation of the TLR2 and TLR4 signalling pathways.

Recently, in a preliminary study the investigators have found that endothelial glycocalyx which is an important part of the vascular barrier and which is intimately linked to the homeostatic functions of the endothelium was altered in APL patients.

Hydroxychloroquine (HCQ) is an antimalarial drug, also used to treat rheumatic diseases such as SLE. There is experimental evidence to suggest a direct role of hydroxychloroquine on the pathophysiology of APS: it directly reduces the binding of antibodies on the phospholipid bilayers, protects the annexin A5 anticoagulant shield and it reverses platelet adhesion induced by aPL.

Furthermore it is known to decrease the expression of lysosomal TLRs, but also extra lysosomal TLR2 and TLR4.

The aim of this study is to investigate whether treatment with hydroxychloroquine modulates vascular endothelial function in patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who fulfilled Sidney criteria for APS (antiphospholipid Syndrome
* Women of childbearing potential must have a contraceptive method
* Written informed consent
* no severe, progressive, or uncontrolled kidney, liver, blood, stomach, lung, heart, or brain disease.

Exclusion Criteria:

* secondary antiphospholipid syndrome
* Pregnancy and breastfeeding
* Patients with a history of severe depression, psychosis, or suicidal ideation
* story of intolerance or contra-indication to hydroxychloroquine, lactose, trinitrin
* Prior use of hydroxychloroquine in the last 6 months
* Chronic heart failure
* atrial fibrillation
* severe pulmonary hypertension
* severe kidney failure clearance < 30ml/mn
* uncontrolled arterial hypertension
* secondary arterial hypertension
* diabetes mellitus diagnosed in the last 3 months
* body mass index > 35
* Patient has been committed to an institution by legal or regulatory order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-05-17 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2020-08-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline flow mediated dilatation of brachial artery | 6 months
  The brachial artery diameter and blood flow are measured by echotracking and Doppler before and just after and ischemic test. Result expressed in percentage of diameter variation.

SECONDARY OUTCOMES:
change from baseline in endothelial glycocalyx thickness | 6 months
  indirect measure of the glycocalyx thickness by using sublingual SDF (sidestream dark field) imaging
change from baseline in oxydative stress | 6 months
  plasma levels of nitrites and TBARS (thiobarbituric acid reactive substance)
change from baseline in systemic inflammation | 6 months
  plasma levels of TNFalpha
change from baseline in coagulation parameter | 6 months
  Tissue factor plasmatic level
change from baseline in plasmatic level in hydroxychloroquine | 6 months
  plasma level of hydroxychloroquine

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien MIRANDA, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France